CLINICAL TRIAL: NCT01449383
Title: Molecular Targets Open for Regulation by the Gut Flora - New Avenues for Improved Diet to Optimize European Health (TORANDO): WP2 Individual Intervention Studies- Effect of Diet on Intestinal Microbiota and Obesity Markers in Adults
Brief Title: Effect of Diet on Intestinal Microbiota and Obesity Markers in Adults
Acronym: TORNADO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Umeå University (Other); Quadram Institute Bioscience (Other); VTT Technical Research Centre of Finland (Other)
Responsible Party: Principal Investigator, Jana Foerster, Jana Foerster, PhD student, German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: KBBE-2007-2-2-07_WP2.4
Record Dates: First submitted 2011-10-05; First posted 2011-10-10 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Intestinal Microbiota; Blood Markers
Keywords: cross over; dietary intervention; fibre; red meat; microbiota

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- low meat high fibre (lmhf) (Active Comparator): consumption of less than 30g red meat per day and at least 40g dietary fibre per day
  Interventions: Dietary Supplement: low meat high fibre
- high meat low fibre (hmlf) (Active Comparator): consumption of 200g red meat and not more than 20g dietary fibre per day
  Interventions: Dietary Supplement: high meat low fibre

INTERVENTIONS:
Dietary Supplement: low meat high fibre — less than 30g red meat and at least 40g dietary fibre per day
  Arms: low meat high fibre (lmhf)
Dietary Supplement: high meat low fibre — at least 200g red meat (pork, beef or other mammals) and not more than 20g dietary fibre per day
  Arms: high meat low fibre (hmlf)

SUMMARY:
This study aims to investigate the direct effect of high amounts of dietary fibre and high amounts of red meat in daily diet on intestinal microbiota, anthropometry and obesity markers in healthy adults.

DETAILED DESCRIPTION:
Human gut microbiota composition and its bacterial pathways are involved in many metabolic processes, including digestion of actually indigestible food components and fat storage. Due to that it may contributes to the developement of obesity being one of the most important risk factors for many chronic diseases. Gut microbiota is under the influence of nutrition, consumption of pro- and prebiotics can promote the growth of certain bacterial strains. In a cross over dietary intervention this work will investigate the effect of defined diets on the intestinal microbiota in 20 healthy adults. The diets contain either high amounts (more than 40g/d) of dietary fibre and low red meat (less than 30g/d) or low amounts (less than 20g/d) of dietary fibre and high amounts of red meat (200g/d). Intervention periods last 3 weeks each interrupted by a 3 weeks wash out period. Examination of participants will happen at the beginning and at the end of both interventions and will contain anthropometry, blood sample, faecal sample, urine sample and saliva sample.

ELIGIBILITY:
Inclusion Criteria:

* age 20 to 60
* obtained informed consent
* willing and able to consume defined diets
* willing and able to collect all intended samples

Exclusion Criteria:

* prevalent chronic disease, i.e. diabetes (type 1 and 2), cardiovascular diseases, cancer
* Antibiotic treatment within the last three month before start of studies
* Prevalent gastrointestinal diseases, disorders and surgeries
* Pregnancy and breastfeeding

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
change in gut microbiota composition | baseline, week 3, 6 and 9

SECONDARY OUTCOMES:
change in anthropometry | baseline, week 3, 6 and 9
  Body height, body weight, circumferences of waist, hip, upper arm and leg, lower leg and the thickness of body folds at waist, back, upper arm and leg, lower leg and thorax depth and width
change in blood markers | baseline, week 3, 6 and 9
  clinical blood count, including Hba1c, gamma-GT, cholesterol, HDL, LDL, Triglycerides, s-creatinin, CRP
change in salivary microbial composition | baseline, week 3, 6 and 9

CONTACTS AND LOCATIONS:
Overall Officials: Jana Foerster, PhD student, Principal Investigator — German Institute of Human Nutrition Potsdam-Rehbruecke

REFERENCES:
- [Derived] Foerster J, Maskarinec G, Reichardt N, Tett A, Narbad A, Blaut M, Boeing H. The influence of whole grain products and red meat on intestinal microbiota composition in normal weight adults: a randomized crossover intervention trial. PLoS One. 2014 Oct 9;9(10):e109606. doi: 10.1371/journal.pone.0109606. eCollection 2014. PMID 25299601